CLINICAL TRIAL: NCT01240395
Title: Mindfulness-based Cognitive Therapy for Individuals With Multiple Chemical Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Danish Research Centre for Chemical Sensitivities (Other)
Responsible Party: Principal Investigator, Christian Riise Hauge, MSc psychology, The Danish Research Centre for Chemical Sensitivities
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBCT-MCS
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Chemical Sensitivity
Keywords: Multiple chemical sensitivities; MCS; Mindfulness-based cognitive therapy; MBCT
MeSH Terms: conditions — Multiple Chemical Sensitivity | interventions — Mindfulness-Based Cognitive Therapy

ARMS (2):
- MBCT intervention (Experimental)
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy (MBCT)
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy (MBCT) — MBCT is partly based on the mindfulness-based stress reduction program (MBSR), developed by Jon Kabat-Zinn and colleagues, and partly on cognitive therapy for depression, the latter influence particularly expressed through the aspect of "decentering", meaning not accepting the content of thoughts as facts and not identifying with the thought. The MBCT programme in this study includes 2½ hours of training once a week for 9 weeks. In addition, participants are encouraged to practice at home for up to 45 min per day, 6 days a week during the entire course.
  Arms: MBCT intervention

SUMMARY:
The objective of this study is to evaluate the effect of mindfulness-based cognitive therapy (MBCT) on physical symptoms attributed to chemical exposures, psychological distress, illness worry, quality of life, and illness perceptions in patients suffering from multiple chemical sensitivity (MCS). Furthermore, a secondary objective is to evaluate whether a possible symptom reduction is mediated by an increased level of mindfulness.

The primary hypothesis is that the self-reported severity of MCS symptoms and the degree to which chemical exposures causes symptoms and the impact on daily life will be significantly improved in the MBCT treatment group as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil Lacour's criteria for Multiple Chemical Sensitivity
* Sign a written informed consent form

Exclusion Criteria:

* A psychotic or bipolar disorder
* An acute psychiatric disorder requiring other treatment
* Suicidal ideations
* Current alcohol or drug abuse
* Previously engaged in a mindfulness programme

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The Quick Environmental Exposure and Sensitivity Inventory (QEESI) | 8 weeks, 1 year follow up
  QEESI is a screening instrument for MCS.

SECONDARY OUTCOMES:
The brief illness perception questionnaire (Brief IPQ) | 8 weeks, 1 year follow up
The Five Facet Mindfulness Questionnaire (FFMQ) | 8 weeks, 1 year follow up
Symptom Check List 92 (SCL-92) | 8 weeks, 1 year follow up
The Perceived Stress Scale (PSS-10) | 8 weeks, 1 year follow up
The World Health Organization Quality of Life (WHOQOL-BREF) | 8 weeks, 1 year follow-up
Rumination-reflection questionnaire (RRQ) | 8 weeks, 1 year follow-up
Self compassion scale short form | 8 weeks, 1 year follow up
The role work functioning index | 8 weeks, 1 year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- The Danish Research Centre for Chemical Sensitivities, Ledreborg Allé 40, 2., Gentofte, Denmark

REFERENCES:
- [Derived] Hauge CR, Bonde PJ, Rasmussen A, Skovbjerg S. Mindfulness-based cognitive therapy for multiple chemical sensitivity: a study protocol for a randomized controlled trial. Trials. 2012 Sep 27;13:179. doi: 10.1186/1745-6215-13-179. PMID 23016822